CLINICAL TRIAL: NCT06640023
Title: The Study in Outpatient Medicine Using Nudges to Improve Sleep: The SOMNUS Trial
Brief Title: The Study in Outpatient Medicine Using Nudges to Improve Sleep
Acronym: SOMNUS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Northwestern Medicine (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jason Doctor, Professor, University of Southern California
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: UP-23-00317; 1R01HL167023-01 (NIH)
Record Dates: First submitted 2024-09-30; First posted 2024-10-15 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Inappropriate Prescribing
Keywords: Sleep Aids, Pharmaceutical; Zolpidem; zaleplon; Eszopiclone; Cognitive Behavioral Therapy; Insomnia; Clinical Decision-Making; Decision Support Systems, Clinical; Economics, Behavioral
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Behavior

STUDY DESIGN:
Intervention Model Description: 2x2
Masking Description: The investigator is masked during data and safety monitoring only.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): Clinicians randomized to this arm receive guideline education prior to the trial.
- Z-drug Default Quantity (Experimental): Clinicians randomized to this arm receive guideline education + 10 pill quantity defaults.
  Interventions: Behavioral: Z-drug Default Quantity
- Redirection + Accountable Justification (Experimental): Clinicians randomized to this arm receive guideline education + alerts requiring justification of orders discordant with guidelines. Justifications are entered in the patient's medical record, and can be viewed by other clinicians.
  Interventions: Behavioral: Redirection + Accountable Justification
- Combined (Experimental): Clinicians randomized to this arm receive guideline education + 10 pill quantity defaults + alerts requiring justification of orders discordant with guidelines. Justifications are entered in the patient's medical record, and can be viewed by other clinicians
  Interventions: Behavioral: Z-drug Default Quantity; Behavioral: Redirection + Accountable Justification

INTERVENTIONS:
Behavioral: Z-drug Default Quantity — For new orders of oral Z-drugs tablets (zolpidem, zolpidem CR, zaleplon, and eszopiclone), the EHR dispense quantity default will be changed to 10 pills with 0 refills for all dosage levels. Dispense quantities for Z-drug reorders and renewals will not be changed.
  Arms: Combined; Z-drug Default Quantity
Behavioral: Redirection + Accountable Justification — For qualifying Z-drug orders, an EHR alert will suggest removing the Z-drug, adding a CBT-I referral, or both. If the alert recommendation is not followed, clinicians will be asked to provide a justification for their decision when the order is signed. The justification will display in the Encounter Report.
  The alert suggestion depends on the recent history of Z-drug prescriptions for a given patient. When a Z-drug is being ordered for patients with 180 days supply of Z-drugs or fewer in the last 365 days, the alert will prompt removal of the Z-drug and addition of a CBT-I referral to the order. When a Z-drug is being ordered for patients with 181 days supply of Z-drugs or more in the last 365 days, the alert will only prompt addition of a CBT-I referral to the order.
  If a CBT-I referral is already in the current order or has been ordered for a patient in the past 180 days, the alert to add a CBT-I referral to the order will not display.
  Arms: Combined; Redirection + Accountable Justification

SUMMARY:
The goal of this clinical trial is to learn if electronic health record (EHR) nudges (changes to the EHR that do not restrict freedom of choice or alter incentives) can reduce Z-drug prescribing in primary care clinics for patients with insomnia. The main questions it aims to answer are:

1. Can Z-drug prescribing be reduced by setting the dispense quantity default of new Z-drug orders in the EHR to 10 pills with 0 refills?
2. Can Z-drug prescribing be reduced by an EHR alert that suggests clinicians remove a Z-drug and/or add an evidence-based behavioral treatment for insomnia, followed by a request to justify their reasoning if the suggestion is not followed?
3. Does combining these two nudges reduce Z-drug prescribing?

Researchers will compare each nudge individually and in combination to an guideline education control group to see if each nudge (separately and in combination) can reduce Z-drug prescribing.

Clinician-participants will:

1. Complete an introductory educational module about treating insomnia and relevant EHR changes.
2. Complete their routine patient visits.
3. Either experience EHR changes when prescribing Z-drugs, including a Z-drug dispense quantity default of 10 pills for new orders, a prompt to remove or justify Z-drug orders, both, or neither.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient primary care clinician at Northwestern Medicine

Exclusion Criteria:

* Clinician participated in pilot study
* Clinician-investigator for this trial
* Visit involves patient with ICD-10 F31.X diagnosis code (bipolar disorder) present in the last year or on active problem list

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 443 (Estimated)
Dates: Start 2024-12-20 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Z-drug pill count | 36 months
  Dose-equivalent Z-drug pill count prescribed at eligible encounters by clinicians from 18 months prior to the intervention start to 18 months after the intervention start.

SECONDARY OUTCOMES:
Z-drug pill count among short-term users | 36 months
  Dose-equivalent Z-drug pill count prescribed at eligible encounters with short-term Z-drug use patients (less than or equal to 180 days of Z-drugs prescribed in last 365 days) by clinicians from 18 months prior to the intervention start to 18 months after the intervention start.
Z-drug pill count among long-term users | 36 months
  Dose-equivalent Z-drug pill count prescribed at eligible encounters of long-term Z-drug use patients (greater than 180 days of Z-drugs prescribed in last 365 days) by clinicians from 18 months prior to the intervention start to 18 months after the intervention start.
CBT-I referrals | 18 months
  Number of patients who are referred to CBT-I from intervention start to 18 months after the intervention start.
CBT-I referrals among short-term users | 18 months
  Number of short-term Z-drug use patients (less than or equal to 180 days of Z-drugs prescribed in last 365 days) who are referred to CBT-I from intervention start to 18 months after the intervention start.
CBT-I referrals among long-term users | 18 months
  Number of long-term Z-drug use patients (greater than 180 days of Z-drugs prescribed in last 365 days) who are referred to CBT-I from intervention start to 18 months after the intervention start.
Monthly Z-drug pill count | 36 months
  Total monthly dose-equivalent Z-drug pill count prescribed by clinicians from 18 months prior to the intervention start to 18 months after the intervention start.
Benzodiazepine pill count | 36 months
  Dose-equivalent benzodiazepine pill count prescribed at eligible encounters by clinicians from 18 months prior to the intervention start to 18 months after the intervention start.
Z-drug guideline discordant duration | 36 months
  Proportion of eligible encounters when patients were prescribed more than 35 Z-drug pills for use within a 5 week period from 18 months prior to the intervention start to 18 months after the intervention start.

OTHER OUTCOMES:
Z-drug pill count at follow-up | 48 months
  Dose-equivalent Z-drug pill count prescribed at eligible encounters by clinicians from 18 months prior to the intervention start to 30 months after the intervention start.
Z-drug pill count at follow-up among short-term users | 48 months
  Dose-equivalent Z-drug pill count prescribed at eligible encounters of short-term Z-drug use patients (less than or equal to 180 days of Z-drugs prescribed in the last 365 days) by clinicians from 18 months prior to the intervention start to 30 months after the intervention start.
Z-drug pill count at follow-up among long-term users | 48 months
  Dose-equivalent Z-drug pill count prescribed at eligible encounters of long-term Z-drug use patients (greater than 180 days of Z-drugs prescribed in the last 365 days) by clinicians from 18 months prior to the intervention start to 30 months after the intervention start.
CBT-I referrals at follow-up | 30 months
  Number of patients who are referred to CBT-I from intervention start to 30 months after the intervention start.
CBT-I referrals at follow-up among short-term users | 30 months
  Number of short-term Z-drug use patients (less than or equal to 180 days of Z-drugs prescribed in last 365 days) who are referred to CBT-I from intervention start to 30 months after the intervention start.
CBT-I referrals at follow-up among long-term users | 30 months
  Number of long-term Z-drug use patients (greater than 180 days of Z-drugs prescribed in last 365 days) who are referred to CBT-I from intervention start to 30 months after the intervention start.
Monthly Z-drug pill count at follow-up | 48 months
  Total monthly dose-equivalent Z-drug pill count prescribed by clinicians from 18 months prior to the intervention start to 30 months after the intervention start.
Benzodiazepine pill count at follow-up | 48 months
  Dose-equivalent benzodiazepine pill count prescribed at eligible encounters by clinicians from 18 months prior to the intervention start to 30 months after the intervention start.
Z-drug guideline discordant duration at follow-up | 48 months
  Proportion of eligible encounters when patients were prescribed more than 35 Z-drug pills for at least 5 consecutive weeks from 18 months prior to the intervention start to 30 months after the intervention start.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Doctor, PhD, Principal Investigator — University of Southern California
Locations (1):
- Northwestern Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data as part of a HIPAA compliant limited data set may be shared with researchers under a signed Data Use Agreement.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be available for one year following study completion date.

REFERENCES:
- [Derived] Cloughesy JN, Linder JA, Knight TK, Persell SD, Sullivan MD, Meeker D, Brown T, Lee JY, Stewart EP, Fox CR, Goldstein NJ, Sumitro RG, Vitiello MV, Mack WJ, Doctor JN. The Study in Outpatient Medicine using Nudges to Improve Sleep (SOMNUS): study protocol for an 18-month factorial, cluster-randomized trial to increase guideline-concordant treatment of insomnia in primary care. Trials. 2025 Dec 23. doi: 10.1186/s13063-025-09385-6. Online ahead of print. PMID 41430294